CLINICAL TRIAL: NCT02265510
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCB052793 in Subjects With Advanced Malignancies
Brief Title: An Open-Label Study of a Novel JAK-inhibitor, INCB052793, Given to Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 52793-101
Expanded Access: NCT03906344 (No longer available)
Record Dates: First submitted 2014-09-29; First posted 2014-10-16 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumors; Advanced Malignancies; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Dexamethasone; carfilzomib; Bortezomib; Lenalidomide; Azacitidine; pomalidomide; parsaclisib; INCB039110; itacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1a: INCB052793 Monotherapy (Experimental)
  Interventions: Drug: INCB052793
- Phase 1b: INCB052793 Combination Therapy (Experimental)
  Interventions: Drug: gemcitabine; Drug: nab-paclitaxel; Drug: dexamethasone; Drug: Carfilzomib; Drug: bortezomib; Drug: lenalidomide; Drug: azacitidine; Drug: INCB052793; Drug: pomalidomide; Drug: INCB050465
- Phase 2: INCB052793 and itacitinib Combination Therapy (Experimental)
  Interventions: Drug: azacitidine; Drug: INCB052793; Drug: INCB039110

INTERVENTIONS:
Drug: INCB052793 — Initial cohort dose of INCB052793 monotherapy at the protocol-specified starting dose, with subsequent cohort escalations based on protocol-specific criteria.
  Arms: Phase 1a: INCB052793 Monotherapy
Drug: gemcitabine — Gemcitabine administered intravenously over 30 minutes at the protocol-specified dose and frequency.
  Other Names: Gemzar®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: nab-paclitaxel — nab-paclitaxel administered intravenously over 30 minutes at the protocol-specified dose and frequency.
  Other Names: Abraxane®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: dexamethasone — Dexamethasone administered orally at the protocol-specified dose and frequency.
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: Carfilzomib — Carfilzomib administered intravenously at the protocol-specified dose and frequency.
  Other Names: Kyprolis®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: bortezomib — Bortezomib administered intravenously or subcutaneously at the protocol-specified dose and frequency.
  Other Names: Velcade®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: lenalidomide — Lenalidomide administered orally at the protocol-specified dose and frequency.
  Other Names: Revlimid®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: azacitidine — Azacitidine administered subcutaneously at the protocol-specified dose and frequency.
  Other Names: Vidaza®
  Arms: Phase 1b: INCB052793 Combination Therapy; Phase 2: INCB052793 and itacitinib Combination Therapy
Drug: INCB052793 — INCB052793 tablets administered orally at the protocol specified dose strength and frequency.
  Arms: Phase 1b: INCB052793 Combination Therapy; Phase 2: INCB052793 and itacitinib Combination Therapy
Drug: pomalidomide — Pomalidomide administered orally at the protocol-specified dose and frequency.
  Other Names: Pomalyst®
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: INCB050465 — INCB050465 tablets administered orally at the protocol specified dose strength and frequency.
  Arms: Phase 1b: INCB052793 Combination Therapy
Drug: INCB039110 — INCB039110 tablets administered orally at the protocol specified dose strength and frequency.
  Other Names: itacitinib
  Arms: Phase 2: INCB052793 and itacitinib Combination Therapy

SUMMARY:
This was a study of INCB052793 given to patients with advanced malignancies that was to be conducted in three phases; Phase 1a (Monotherapy) and Phase 1b (Combination Therapy) and Phase 2 (Combination therapy of INCB052793 with azacitidine and itacitinib with azacitidine). Phase 1 had two parts; a dose escalation (Part 1) and an expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Phase 1a

* Aged 18 years or older
* Histologically or cytologically confirmed solid tumor or hematologic malignancy
* Life expectancy of 12 weeks or longer
* Must have received ≥ 1 prior treatment regimen
* Must not be a candidate for potentially curative or standard of care approved therapy

Phase 1b

* Aged 18 years or older
* Cohort A: Histologically or cytologically confirmed pancreatic adenocarcinoma, triple-negative breast cancer, urothelial cancer with at least 1 measurable or evaluable target lesion
* Cohorts B, C, D, E and G: Histologically confirmed multiple myeloma and measureable/evaluable disease
* Cohort F: Confirmed acute myeloid leukemia or myelodysplastic syndrome
* Cohort H: Individuals diagnosed with lymphoma
* Prior therapy:

  * Cohort A: No more than 1 prior chemotherapy regimen for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy)
  * Cohorts B, C, D, E and G: Must have relapsed from or have been refractory to ≥ 2 prior treatment regimens
  * Cohort F: May have received any number of prior treatment regimens or be treatment-naïve
  * Cohort H: Must have relapsed from or have been refractory to available treatments

Phase 2

* Aged 18 years or older
* Cohorts I and J: Confirmed acute myeloid leukemia or high risk myelodysplastic syndrome
* Prior therapy:

  * Cohorts I and J: Must have failed prior therapy with a hypomethylating agent (HMA)

Exclusion Criteria:

* Prior receipt of a JAK1 inhibitor (Phase 1a only)
* Known active central nervous system metastases and/or carcinomatous meningitis
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Any known contraindications to the use of gemcitabine, nab-paclitaxel, dexamethasone, carfilzomib, bortezomib, lenalidomide, azacitidine, pomalidomide or PI3Kδ inhibitor (Phase 1b and Phase 2 only, as appropriate to treatment cohort)
* Known human immunodeficiency virus infection, or evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterine Asatiani, M.D., Study Director — Incyte Corporation
Locations (14):
- United States (14):
  - Birmingham, Alabama
  - West Hollywood, California
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Hackensack, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Portland, Oregon
  - Greenville, South Carolina
  - Site 2, Nashville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in United States from 10 September 2014 to 27 February 2019. This study was prematurely terminated due to lack of efficacy.
Pre-assignment Details: Participants with advanced malignancies,acute myeloid leukemia(AML),high-risk myelodysplastic syndrome(MDS)who failed prior therapy with hypomethylating agents(HMA)enrolled to dose escalation(Part 1),expansion(Part 2) of INCB052793 monotherapy and combination therapy cohorts.CohortsA,C,D,E,G,H had no enrollment at the time of premature termination.
Groups:
- Phase 1a TGA - INCB052793 15 mg: INCB052793 15 mg tablet, orally (PO), once daily (QD) in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGA - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21day cycles until they met treatment discontinuation criteria
- Phase 1a TGA - INCB052793 35 mg: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21day cycles until they met treatment discontinuation criteria.
- Phase 1a TGA - INCB052793 50 mg: INCB052793 50 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGA - INCB052793 75 mg: INCB052793 75 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGA - INCB052793 100 mg: INCB052793 100 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGB - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21day cycles until they met treatment discontinuation criteria.
- Phase 1a TGB - INCB052793 35 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGB - INCB052793 50 mg: INCB052793 50 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria
- Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with multiple myeloma (MM) in continuous 21 day cycles until they met treatment discontinuation criteria plus Dexamethasone 40 mg, PO, weekly for each 21-day cycle.
- Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with acute myeloid leukemia (AML)/ myelodysplastic syndrome (MDS) in continuous 21day cycles until they met treatment discontinuation criteria plus Azacitidine 75 mg/m^2, subcutaneous (SC) injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Hase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with AML/MDS in continuous 21 day cycles until they met treatment discontinuation criteria Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 28-day cycle.
- Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with hypomethylating agent-refractory (HMA)-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2: Itacitinib 300 mg sustained-release tablet, PO, QD in the fasted state in participants with HMA-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle
Period: Overall Study
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1a TGB - INCB052793 25 mg | Phase 1a TGB - INCB052793 35 mg | Phase 1a TGB - INCB052793 50 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Hase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
Started | 3 | 3 | 6 | 4 | 3 | 6 | 3 | 4 | 4 | 7 | 5 | 16 | 9 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 4 | 3 | 6 | 3 | 4 | 4 | 7 | 5 | 16 | 9 | 10
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 2 | 2 | 1 | 3 | 2 | 1 | 3 | 3 | 4 | 12 | 7 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The safety evaluable population included all subjects enrolled in the study who receivedat least 1 dose of study treatment.
Groups:
- Phase 1a TGA - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGA - INCB052793 35 mg: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria
- Phase 1a TGB - INCB052793 25 mg; Phase 1a TGB - INCB052793 35 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with acute myeloid leukemia (AML)/ myelodysplastic syndrome (MDS) in continuous 21 day cycles until they met treatment discontinuation criteria plus Azacitidine 75 mg/m^2, subcutaneous (SC) injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with AML/MDS in continuous 21 day cycles until they met treatment discontinuation criteria Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle
- • Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2: Itacitinib 300 mg sustained-release tablet, PO, QD in the fasted state in participants with HMA-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1a TGB - INCB052793 25 mg | Phase 1a TGB - INCB052793 35 mg | Phase 1a TGB - INCB052793 50 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 | • Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 3 | 6 | 3 | 4 | 4 | 7 | 5 | 16 | 9 | 10 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.08) | 59.0 (9.85) | 57.0 (13.19) | 54.5 (13.40) | 46.0 (15.13) | 63.0 (10.77) | 60.3 (6.66) | 58.5 (6.45) | 56.3 (3.69) | 60.3 (13.84) | 62.8 (14.17) | 64.4 (15.47) | 70.4 (5.64) | 71.2 (8.50) | 62.6 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 2 | 4 | 1 | 0 | 1 | 0 | 3 | 7 | 2 | 2 | 29
  Male | 2 | 1 | 4 | 2 | 1 | 2 | 2 | 4 | 3 | 7 | 2 | 9 | 7 | 8 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 | 3 | 5 | 2 | 2 | 5 | 2 | 3 | 4 | 5 | 5 | 14 | 9 | 8 | 70
  Black/African-American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 8
  American-Indian/Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 2 | 3 | 6 | 4 | 2 | 6 | 2 | 3 | 4 | 6 | 5 | 16 | 9 | 10 | 78
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a and 1b: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a subject administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization. A TEAE was defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last dose of study drug.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (Up to approximately 3.4 years)
Population: Safety evaluable population included all participants exposed to ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1a TGA - INCB052793 25 mg; Phase 1a TGB - INCB052793 25 mg; Phase 1a TGB - INCB052793 35 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria.
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1a TGB - INCB052793 25 mg | Phase 1a TGB - INCB052793 35 mg | Phase 1a TGB - INCB052793 50 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 3 | 6 | 3 | 4 | 4 | 7 | 5 | 16
Participants
  TEAE | 3 | 3 | 6 | 4 | 3 | 6 | 3 | 4 | 4 | 7 | 5 | 16
  SAE | 0 | 1 | 0 | 2 | 3 | 2 | 1 | 2 | 2 | 5 | 4 | 14
Statistical Analysis 1: Comparison: Phase 1a TGA - INCB052793 15 mg vs Phase 1a TGA - INCB052793 25 mg vs Phase 1a TGA - INCB052793 35 mg vs Phase 1a TGA - INCB052793 50 mg vs Phase 1a TGA - INCB052793 75 mg vs Phase 1a TGA - INCB052793 100 mg vs Phase 1a TGB - INCB052793 25 mg vs Phase 1a TGB - INCB052793 35 mg vs Phase 1a TGB - INCB052793 50 mg vs Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg vs Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 vs Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2; Test type: Other — Descriptive Statistics; The analysis of the primary endpoint was descriptive i.e. no statistical hypothesis test was performed

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) in Hematological Malignancies
Description: ORR is defined as the proportion of participants who achieved complete response (CR), CR with incomplete hematologic recovery (CRi), partial response (PR), or hematologic improvement (HI), using the IWG response criteria.
Time Frame: Baseline through end of study (Up to approximately 4.5 years)
Population: Efficacy evaluable population included all participants exposed to ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Cohort I-INCB052793 +Azacytidine (AML): INCB052793 35 mg tablet, PO, QD in the fasted state in participants with HMA-refractory AML in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Phase 2 Cohort I-INCB052793 +Azacytidine (MDS): INCB052793 35 mg tablet, PO, QD in the fasted state in participants with high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Phase 2 Cohort J-Itacitinib +Azacitidine (AML): Itacitinib 300 mg sustained-release tablet, PO, QD in the fasted state in participants with HMA-refractory AML in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
- Phase 2 Cohort J-Itacitinib +Azacitidine (MDS): Itacitinib 300 mg sustained-release tablet, PO, QD in the fasted state in participants with high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle .
Arm/Group | Phase 2 Cohort I-INCB052793 +Azacytidine (AML) | Phase 2 Cohort I-INCB052793 +Azacytidine (MDS) | Phase 2 Cohort J-Itacitinib +Azacitidine (AML) | Phase 2 Cohort J-Itacitinib +Azacitidine (MDS)
Number analyzed (Participants) | 6 | 3 | 8 | 2
Participants | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Phase 2 Cohort I-INCB052793 +Azacytidine (AML) vs Phase 2 Cohort I-INCB052793 +Azacytidine (MDS) vs Phase 2 Cohort J-Itacitinib +Azacitidine (AML) vs Phase 2 Cohort J-Itacitinib +Azacitidine (MDS); Test type: Other; Confidence Intervals for ORR were calculated based on the exact method for binomial distributions. There were no comparison between treatment groups

3. Secondary Outcome: Phase 1A and 1B: Percentage of Participants With Response as Determined by Investigator's Assessment
Description: Response rate is defined as the percentage of participants who achieved best overall response (BOR) as determined by IWG response criteria of investigator's assessment. A participant was considered an objective responder based on the following- Solid tumors: participant had a best overall response (BOR) of CR or PR, Lymphoma: participant had a BOR of complete radiologic response/complete metabolic response or partial remission/partial metabolic response, AML: participant had a BOR of CR, CRi, morphological leukemia-free state (MLFS), or PR, MDS: participant had a BOR of CR, PR, or marrow CR, MDS/myeloproliferative neoplasm (MPN): participant had a BOR of CR, PR, or marrow response, MM: participant had a BOR of stringent CR, CR, very good PR, PR, or MR. Subjects are combined by tumor type for this analysis.
Time Frame: Baseline through end of study (Up to approximately 4.5 years)
Population: Efficacy evaluable population included all participants exposed to ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1a TGA - INCB052793 in Solid Tumors: INCB052793 tablet, orally (PO), once daily (QD) in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1a TGB - INCB052793 in Lymphoma; Phase 1a TGB - INCB052793 in MDS/MPN; Phase 1a TGB - INCB052793 in MM: INCB052793 tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria.
- Phase 1b Cohort B - INCB052793 + Dexamethasone in MM: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with multiple myeloma (MM) in continuous 21 day cycles until they met treatment discontinuation criteria plus Dexamethasone 40 mg, PO, weekly for each 21-day cycle.
- Phase 1b Cohort F-INCB052793 +Azacytidine in AML; Phase 1b Cohort F-INCB052793 +Azacytidine in MDS; Phase 1b Cohort F-INCB052793 +Azacytidine in MDS/MPN: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with acute myeloid leukemia (AML)/ myelodysplastic syndrome (MDS) in continuous 21 day cycles until they met treatment discontinuation criteria plus Azacitidine 75 mg/m^2, subcutaneous (SC) injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle.
Arm/Group | Phase 1a TGA - INCB052793 in Solid Tumors | Phase 1a TGB - INCB052793 in Lymphoma | Phase 1a TGB - INCB052793 in MDS/MPN | Phase 1a TGB - INCB052793 in MM | Phase 1b Cohort B - INCB052793 + Dexamethasone in MM | Phase 1b Cohort F-INCB052793 +Azacytidine in AML | Phase 1b Cohort F-INCB052793 +Azacytidine in MDS | Phase 1b Cohort F-INCB052793 +Azacytidine in MDS/MPN
Number analyzed (Participants) | 25 | 4 | 4 | 3 | 7 | 12 | 7 | 2
Participants | 0 | 0 | 1 | 0 | 2 | 4 | 3 | 2
Statistical Analysis 1: Comparison: Phase 1a TGA - INCB052793 in Solid Tumors vs Phase 1a TGB - INCB052793 in Lymphoma vs Phase 1a TGB - INCB052793 in MDS/MPN vs Phase 1a TGB - INCB052793 in MM vs Phase 1b Cohort B - INCB052793 + Dexamethasone in MM vs Phase 1b Cohort F-INCB052793 +Azacytidine in AML vs Phase 1b Cohort F-INCB052793 +Azacytidine in MDS vs Phase 1b Cohort F-INCB052793 +Azacytidine in MDS/MPN; Test type: Other; Confidence Intervals for response were calculated based on the exact method for binomial distributions. There were no comparison between treatment groups

4. Secondary Outcome: Phase 2: Number of Participants With at Least One TEAE and SAE
Description: as for outcome 1
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (Up to approximately 1.3 years)
Population: Safety evaluable population included all participants exposed to ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9 | 10
Participants
  TEAE | 9 | 10
  SAE | 7 | 8
Statistical Analysis 1: Comparison: Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 vs Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

5. Secondary Outcome: Phase 1a, 1b, and Phase 2: Cmax: Maximum Observed Plasma Concentration for INCB052793
Description: Cmax is defined as the maximum observed plasma concentration measured at steady state (Day 15). For PK analyses subjects in TGA and TGB are combined by dosage group because only 3 subjects were enrolled in each dose group in TGB and 4 subject for first dose in TGB 50 mg.
Time Frame: Cycle 1, Day 15: predose and 0.5, 1, 2, 4, 6 hours postdose in Phase 1a; 0 (predose), 0.08, 0.5, 1, 2, 4, 6 and 8 hours postdose in Phase 1b and Phase 2
Population: The PK evaluable population includes all subjects who received at least 1 dose of study treatment and provided serial samples for PK analysis
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Phase 1a TGA - INCB052793 15 mg: INCB052793 15 mg tablet, orally (PO), once daily (QD) in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 78.3 days ).
- Phase 1a TGA - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 96.3 days).
- Phase 1a TGA - INCB052793 35 mg: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 80.3 days).
- Phase 1a TGA - INCB052793 50 mg: INCB052793 50 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 46.5 days).
- Phase 1a TGA - INCB052793 75 mg: INCB052793 75 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 459.0 days).
- Phase 1a TGA - INCB052793 100 mg: INCB052793 100 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 44.0 days).
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 3 | 3 | 6 | 6 | 15 | 8
nM | 522 (126) | 1110 (324) | 1120 (543) | 2050 (1070) | 1840 (563) | 2890 (1690) | 928 (263) | 1270 (856) | 1480 (588) | 1610 (745)
Statistical Analysis 1: Comparison: Phase 1a TGA - INCB052793 15 mg vs Phase 1a TGA - INCB052793 25 mg vs Phase 1a TGA - INCB052793 35 mg vs Phase 1a TGA - INCB052793 50 mg vs Phase 1a TGA - INCB052793 75 mg vs Phase 1a TGA - INCB052793 100 mg vs Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg vs Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 vs Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 vs Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

6. Secondary Outcome: Phase 1a, 1b, and Phase 2: Tmax: Time to Maximum Plasma Concentration for INCB052793
Description: Tmax is the time to maximum (peak) observed plasma drug concentration. Summary of Steady-State, Day 15, was evaluated by dosing regimen. For PK analyses subjects in TGA and TGB are combined by dosage group because only 3 subjects were enrolled in each dose group in TGB and 4 subject for first dose in TGB 50 mg.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 3 | 3 | 6 | 6 | 15 | 8
hours (hr) | 1.1 [0.48 to 2.0] | 0.76 [0.47 to 2.0] | 2.0 [0.50 to 4.0] | 1.1 [1.0 to 2.1] | 2.2 [1.1 to 4.0] | 2.0 [0.43 to 2.1] | 1.0 [0.43 to 2.0] | 1.1 [0.58 to 7.7] | 1.1 [0.47 to 2.1] | 0.51 [0.33 to 2.1]
Statistical Analysis 1: Comparison: Phase 1a TGA - INCB052793 15 mg vs Phase 1a TGA - INCB052793 25 mg vs Phase 1a TGA - INCB052793 35 mg vs Phase 1a TGA - INCB052793 50 mg vs Phase 1a TGA - INCB052793 75 mg vs Phase 1a TGA - INCB052793 100 mg vs Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg vs Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 vs Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 vs Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

7. Secondary Outcome: Phase 1a, 1b, and Phase 2: AUC0-τ: Area Under the Plasma Concentration-time Curve Over Dosing Interval for INCB052793
Description: AUC0-τ is the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t measured at steady state (Day 15). For PK analyses subjects in TGA and TGB are combined by dosage group because only 3 subjects were enrolled in each dose group in TGB and 4 subject for first dose in TGB 50 mg.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nM*hr
Groups:
- Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with multiple myeloma (MM) in continuous 21 day cycles until they met treatment discontinuation criteria plus Dexamethasone 40 mg, PO, weekly for each 21-day cycle .
- Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with hypomethylating agent-refractory (HMA)-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 21-day cycle .
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 3 | 3 | 6 | 6 | 15 | 8
nM*hr | 4750 (1380) | 9170 (4290) | 8430 (2520) | 14700 (6670) | 18300 (10600) | 27800 (12300) | 6390 (1690) | 9580 (6710) | 10200 (5260) | 9380 (4390)
Statistical Analysis 1: Comparison: Phase 1a TGA - INCB052793 15 mg vs Phase 1a TGA - INCB052793 25 mg vs Phase 1a TGA - INCB052793 35 mg vs Phase 1a TGA - INCB052793 50 mg vs Phase 1a TGA - INCB052793 75 mg vs Phase 1a TGA - INCB052793 100 mg vs Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg vs Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 vs Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 vs Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

8. Secondary Outcome: Phase 1a, 1b, and Phase 2: Cmax: Maximum Observed Plasma Concentration of Itacitinib
Description: Cmax is defined as the maximum observed plasma concentration measured at steady state (Day 15).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9
nM | 1310 (638)
Statistical Analysis 1: Comparison: Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

9. Secondary Outcome: Phase 1a, 1b, and Phase 2: Tmax: Time to Maximum Plasma Concentration for Itacitinib
Description: Tmax is the time to maximum (peak) observed plasma drug concentration.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9
hr | 3.5 [1.0 to 8.0]
Statistical Analysis 1: Comparison: Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

10. Secondary Outcome: Phase 1a, 1b, and Phase 2: AUC0-τ: Area Under the Plasma Concentration-time Curve Over Dosing Interval for Itacitinib
Description: AUC0-τ is the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t measured at steady state (Day 15).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 9
nM*hr | 9870 (7350)
Statistical Analysis 1: Comparison: Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

11. Secondary Outcome: Phase 1a, Part 2: Cmax: Maximum Observed Plasma Concentration for INCB052793
Description: Cmax is defined as the maximum observed plasma concentration measured at Day 1.
Time Frame: Cycle 1, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Groups:
- Phase 1a Part 2 Expasion Cohort- INCB052793: INCB052793 35 mg tablet in combination with Azacitidine or Itacitinib 300mg in combination with Azacitidine
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Phase 1a Part 2 Expasion Cohort- INCB052793; Test type: Other; The analysis of the endpoint was descriptive i.e. no statistical hypothesis test was performed

12. Secondary Outcome: Phase 1a, Part 2: Tmax: Time to Maximum Plasma Concentration for INCB052793
Description: Tmax is the time to maximum (peak) observed plasma drug concentration.
Time Frame: Cycle 1, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 1a, Part 2: AUC[0-t]: Area Under the Plasma Concentration-Time Curve From Time 0 To the Last Measurable Concentration at Time t
Description: AUC0-t is the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t.
Time Frame: Cycle 1, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 1a, Part 2: Cmax: Maximum Observed Plasma Concentration for INCB052793
Description: Cmax is defined as the maximum observed plasma concentration measured at steady state (Day 15).
Time Frame: Cycle 1, Day 15
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1a, Part 2: Cmin: Minimum Observed Plasma Concentration Over the Dose Interval
Description: Minimum observed plasma concentration measured at steady state (Day 15).
Time Frame: Cycle 1, Day 15
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 1a, Part 2: Tmax: Time to Maximum Plasma Concentration for INCB052793
Description: Tmax is the time to maximum (peak) observed plasma drug concentration.
Time Frame: Cycle 1, Day 15
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 1a, Part 2: AUC[0-t]: Area Under the Plasma Concentration-Time Curve From Time 0 To the Last Measurable Concentration at Time
Description: AUC0-t is the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t measured at steady state (Day 15).
Time Frame: Cycle 1, Day 15
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase 1a, Part 2: AUC0-τ: Area Under the Plasma Concentration-time Curve Over Dosing Interval for INCB052793
Description: AUC0-τ is the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t.
Time Frame: Cycle 1, Day 15
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase 1a, Part 2: Cmax: Maximum Observed Plasma Concentration for INCB052793
Description: Cmax is defined as the maximum observed plasma concentration measured at cycle 2 Day 1.
Time Frame: Cycle 2, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

20. Secondary Outcome: Phase 1a, Part 2: Cmin: Minimum Observed Plasma Concentration Over the Dose Interval
Description: Cmin is defined as the minimal observed plasma concentration measured at cycle 2 Day 1
Time Frame: Cycle 2, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

21. Secondary Outcome: Phase 1a, Part 2: Tmax: Time to Maximum Plasma Concentration for INCB052793
Description: Tmax is the time to maximum (peak) observed plasma drug concentration.
Time Frame: Cycle 2, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

22. Secondary Outcome: Phase 1a, Part 2: AUC[0-t]: Area Under the Plasma Concentration-Time Curve From Time 0 To the Last Measurable Concentration at Time
Description: as for outcome 13
Time Frame: Cycle 2, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase 1a, Part 2: AUC0-τ: Area Under the Plasma Concentration-time Curve Over Dosing Interval for INCB052793
Description: as for outcome 18
Time Frame: Cycle 2, Day 1
Population: Data was not collected as no participants were enrolled in Part 2 of the study
Arm/Group | Phase 1a Part 2 Expasion Cohort- INCB052793
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30-35 days after last dose of study drug (Up to approximately 3.4 years)
Groups:
- Phase 1a TGA - INCB052793 15 mg: INCB052793 15 mg tablet, orally (PO), once daily (QD) in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 78.3 days ).
- Phase 1a TGA - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced or metastatic solid tumors treated in continuous 21day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 96.3 days).
- Phase 1a TGB - INCB052793 25 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 248.7 days).
- Phase 1a TGB - INCB052793 35 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 342.8 days).
- Phase 1a TGB - INCB052793 50 mg: INCB052793 50 mg tablet, PO, QD in the fasted state in participants with advanced hematologic malignancies treated in continuous 21 day cycles until they met treatment discontinuation criteria (Up to mean duration of exposure of approximately 76.3 days).
- Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with multiple myeloma (MM) in continuous 21 day cycles until they met treatment discontinuation criteria plus Dexamethasone 40 mg, PO, weekly for each 28-day cycle (Up to mean duration of exposure of approximately 53.6 days).
- Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2: INCB052793 25 mg tablet, PO, QD in the fasted state in participants with acute myeloid leukemia (AML)/ myelodysplastic syndrome (MDS) in continuous 21 day cycles until they met treatment discontinuation criteria plus Azacitidine 75 mg/m^2, subcutaneous (SC) injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 28-day cycle (Up to mean duration of exposure of approximately 151.2 days).
- Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with AML/MDS in continuous 21 day cycles until they met treatment discontinuation criteria Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 28-day cycle (Up to mean duration of exposure of approximately 142.1 days).
- Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2: INCB052793 35 mg tablet, PO, QD in the fasted state in participants with hypomethylating agent-refractory (HMA)-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 28-day cycle (Up to mean duration of exposure of approximately 86.2 days).
- Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2: Itacitinib 300 mg sustained-release tablet, PO, QD in the fasted state in participants with HMA-refractory AML and high-risk MDS in continuous 21 day cycles until they met treatment discontinuation criteria. Azacitidine 75 mg/m^2, SC injection for 5 days, then no treatment for 2 days, then 75 mg/m^2 for 2 days for each 28-day cycle (Up to mean duration of exposure of approximately 143 days).
Arm/Group | Phase 1a TGA - INCB052793 15 mg | Phase 1a TGA - INCB052793 25 mg | Phase 1a TGA - INCB052793 35 mg | Phase 1a TGA - INCB052793 50 mg | Phase 1a TGA - INCB052793 75 mg | Phase 1a TGA - INCB052793 100 mg | Phase 1a TGB - INCB052793 25 mg | Phase 1a TGB - INCB052793 35 mg | Phase 1a TGB - INCB052793 50 mg | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 2/6 | 2/4 | 1/3 | 3/6 | 2/3 | 1/4 | 3/4 | 3/7 | 4/5 | 12/16 | 7/9 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/6 | 2/4 | 3/3 | 2/6 | 1/3 | 2/4 | 2/4 | 5/7 | 4/5 | 14/16 | 7/9 | 8/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 4/4 | 3/3 | 6/6 | 3/3 | 4/4 | 4/4 | 7/7 | 5/5 | 16/16 | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1a TGA - INCB052793 15 mg (N=3) | Phase 1a TGA - INCB052793 25 mg (N=3) | Phase 1a TGA - INCB052793 35 mg (N=6) | Phase 1a TGA - INCB052793 50 mg (N=4) | Phase 1a TGA - INCB052793 75 mg (N=3) | Phase 1a TGA - INCB052793 100 mg (N=6) | Phase 1a TGB - INCB052793 25 mg (N=3) | Phase 1a TGB - INCB052793 35 mg (N=4) | Phase 1a TGB - INCB052793 50 mg (N=4) | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg (N=7) | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 (N=5) | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 (N=16) | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 (N=9) | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2 (N=10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 9 | 3 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a TGA - INCB052793 15 mg (N=3) | Phase 1a TGA - INCB052793 25 mg (N=3) | Phase 1a TGA - INCB052793 35 mg (N=6) | Phase 1a TGA - INCB052793 50 mg (N=4) | Phase 1a TGA - INCB052793 75 mg (N=3) | Phase 1a TGA - INCB052793 100 mg (N=6) | Phase 1a TGB - INCB052793 25 mg (N=3) | Phase 1a TGB - INCB052793 35 mg (N=4) | Phase 1a TGB - INCB052793 50 mg (N=4) | Phase 1b Cohort B - INCB052793 25 mg + Dexamethasone 40 mg (N=7) | Phase 1b Cohort F - INCB052793 25 mg + Azacytidine 75 mg/m^2 (N=5) | Phase 1b Cohort F - INCB052793 35 mg + Azacytidine 75 mg/m^2 (N=16) | Phase 2 Cohort I - INCB052793 35 mg + Azacytidine 75 mg/m^2 (N=9) | Phase 2 Cohort J - Itacitinib 300 mg + Azacitidine 75 mg/m^2 (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 3 | 2 | 10 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 4 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 2 | 1 | 4 | 1 | 7 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 3 | 8 | 4 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 5 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 7 | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 5 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 1 | 3 | 0 | 2
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 3
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 2 | 2 | 3 | 0 | 0 | 3 | 2 | 3 | 8 | 2 | 5
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 4 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 0 | 2 | 3 | 1 | 2 | 0 | 3 | 1 | 5 | 3 | 2
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 6 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood iron increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Human papilloma virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 3 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 4 | 1 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 5 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 3 | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 5 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT02265510/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT02265510/SAP_001.pdf